CLINICAL TRIAL: NCT01332422
Title: Special Drug Use Investigation for ADOAIR Metered-dose Inhaler (Pediatric)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113405
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric patients prescribed ADOAIR: Pediatric patients with asthma prescribed ADOAIR during study period
  Interventions: Drug: Salmeterol and Fluticasone

INTERVENTIONS:
Drug: Salmeterol and Fluticasone — Collection of safety data

SUMMARY:
To investigate possible problems or questions in safety and efficacy of ADOAIR 100 DISKUS and ADOAIR 50 AEROSOL 120 in Japanese pediatric patients with bronchial asthma for a long term under the practical use conditions. In this special drug use investigation, the following items shall be handled as the priority investigation items for information collection.

1. Systemic effects accompanying steroid administration; influences on adrenocortical function, influences on bone metabolisms (fracture, osteoporosis, etc.), cataract, glaucoma
2. Events related to nervous system, musculoskeletal system and circulatory system; tremor, headache, cramp, tachycardia, etc.

ELIGIBILITY:
Inclusion Criteria:

* ADOAIR must be used for the first time
* ADOAIR used for a long-term

Exclusion Criteria:

* Patients with hypersensitivity to salmeterol and fluticasone
* Patients with infection which salmeterol and fluticasone is not effective
* Patients with deep mycosis

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Japanese pediatric patients (aged < 15 years) who diagnosed as having bronchial asthma for which the indication of ADOAIR has been approved and who are using ADOAIR for the first time and expected for a long-term use.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy for a long term under the practical use conditions. As the priority investigation items, (1)Systemic effects accompanying steroid administration (2) Events related to nervous system, musculoskeletal system and circulatory systems | One year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline